CLINICAL TRIAL: NCT05816278
Title: The Association Between Anemia (Hemoglobin Level) and Cardiomegaly Based On Chest Radiograph and Echocardiography
Brief Title: The Association Between Anemia and Cardiomegaly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Putri Amelia, dr. Putri Amelia, M.Ked (Ped), Sp.A(K), Universitas Sumatera Utara
Other Study IDs: 001
Record Dates: First submitted 2023-04-02; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Anemia in Children; Cardiomegaly
MeSH Terms: conditions — Cardiomegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Anemia is one of the major global problems that continues to this day. According to World Health Organization (WHO) data, anemia is found in 1.62 billion people or equivalent to 24.8% of the world's population while, the prevalence of anemia in children under 6 years of age in Indonesia reached 38.4%. Anemia, if undiagnosed or untreated for a long period of time can lead to multiorgan failure. The cardiovascular system is the most commonly affected system in chronic anemia. Between one-third and two-thirds of patients with severe anemia have cardiomegaly and this will return to normal within a few weeks after the anemia is well managed. This abnormality can be evaluated on chest radiograph or echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Anemia patients aging maximum 18 years old
* Anemia patients who had undergone chest radiograph and echocardiography

Exclusion Criteria:

* Anemia patients who had undergone definitive surgery
* Anemia patients who had took iron supplementation in the last 3 months
* Anemia patients who had other anemic conditions such as chronic kidney disease or hemolytic anemia

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children diagnosed with anemia; whether from the pediatric ward and pediatric cardiology outpatient clinic
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Anemia | April 2023 - September 2023
  Diagnosis of anemia based on Hb levels according to WHO classification
Cardiomegaly | April 2023 - September 2023
  Diagnosis of cardiomegaly based on chest radiograph and echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Sumatera Utara, Medan, North Sumatera, Indonesia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05816278/Prot_SAP_000.pdf